CLINICAL TRIAL: NCT03043391
Title: Phase Ib Study of Oncolytic Polio/Rhinovirus Recombinant Against Recurrent Malignant Glioma in Children
Brief Title: Phase 1b Study PVSRIPO for Recurrent Malignant Glioma in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Istari Oncology, Inc. (Industry)
Collaborators: Solving Kids' Cancer (Other); The Andrew McDonough B+ Foundation (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00071228
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2022-06

CONDITIONS: Malignant Glioma; Anaplastic Astrocytoma; Anaplastic Oligoastrocytoma; Anaplastic Oligodendroglioma; Glioblastoma; Gliosarcoma; Atypical Teratoid/Rhabdoid Tumor of Brain; Medulloblastoma; Ependymoma; Pleomorphic Xanthoastrocytoma of Brain; Embryonal Tumor of Brain
Keywords: Pediatric Malignant Glioma; PVSRIPO; Pro00071228; Eric Thompson; Darell Bigner; Oncolytic Poliovirus; Daniel Landi
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Medulloblastoma; Ependymoma

STUDY DESIGN:
Intervention Model Description: Phase Ib study to evaluate feasibility, safety, and preliminary evidence of efficacy of the optimal adult dose in a pediatric population
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Polio/Rhinovirus Recombinant (PVSRIPO) (Experimental): PVSRIPO is an altered form of the live polio vaccine. It was produced by removing a piece of the virus and replacing it with a piece from a common cold virus. This was done to make sure PVSRIPO cannot cause polio even when injected into the brain.
  Interventions: Biological: Polio/Rhinovirus Recombinant (PVSRIPO)

INTERVENTIONS:
Biological: Polio/Rhinovirus Recombinant (PVSRIPO) — PVSRIPO will be delivered intratumorally by convection-enhanced delivery (CED) using an intracerebral catheter placed within the enhancing portion of the tumor. A stereotactic biopsy will be performed prior to virus administration. Immediately following the stereotactically-guided tumor biopsy, a catheter will be implanted in the operating room at a site the same or different from that used for the biopsy using sterile techniques under general anesthesia. The entire volume of PVSRIPO to be delivered will be pre-loaded into a syringe by the investigational pharmacist and connected to the catheter under sterile conditions in the Pediatric Intensive Care Unit (PICU) just prior to beginning of infusion.

SUMMARY:
The purpose of the study is to confirm the safety of the selected dose and potential toxicity of oncolytic poliovirus (PV) immunotherapy with PVSRIPO for pediatric patients with recurrent WHO grade III or IV malignant glioma, but evidence for efficacy will also be sought. The primary objective is to confirm the safety of the selected dose of PVSRIPO when delivered intracerebrally by convection-enhanced delivery (CED) in children with recurrent WHO Grade III malignant glioma (anaplastic astrocytoma, anaplastic oligoastrocytoma, anaplastic oligodendroglioma, anaplastic pleomorphic xanthoastrocytoma) or WHO Grade IV malignant glioma (glioblastoma, gliosarcoma). A secondary objective is to estimate overall survival (OS) in this population.

DETAILED DESCRIPTION:
PVSRIPO will be delivered intratumorally by CED using an intracerebral catheter placed within the enhancing portion of the tumor. The population group are patients with recurrent WHO grade III or IV malignant glioma who are aged 12 through 21 years old. After a single dose of PVSRIPO, subjects will return for periodic visits to monitor tumor status, adverse events, and changes in blood immune profiles. A maximum of 12 pediatric patients will be treated with PVSRIPO, and then carefully monitored for safety for at least a year after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a recurrent supratentorial WHO Grade III malignant glioma (anaplastic astrocytoma, anaplastic oligoastrocytoma, anaplastic oligodendroglioma, anaplastic pleomorphic xanthoastrocytoma, ependymoma) or WHO Grade IV malignant glioma, medulloblastoma, or atypical teratoid/rhabdoid tumor (ATRT) based on imaging studies with measurable disease (≥ 1 cm and ≤ 5.5 cm). The prior histopathology must be consistent with a World Health Organization (WHO) Grade III or IV malignant tumor confirmed by the study pathologist, Roger McLendon, or his designee.
* There is no standard of care treatment for children with Grade III/IV gliomas; however, patients must have received some form of definitive treatment, i.e., standard therapy with known clinical benefit, for their initial diagnosis prior to their recurrence/progression. Definitive treatment includes maximal safe resection (if possible) and radiation therapy with or without chemotherapy. (Please note that patients who are unable to receive radiation therapy due to genetic disorders that put them at significant risk for radiation-induced secondary malignancies (i.e., Gorlin's syndrome or NF1 mutation) are still eligible to participate).
* Due to the potential implications of the treatment on the developing CNS, all patients must be ≥ 12 years of age and ≤ 21 years of age at the time of entry into the study.
* The patient must have a Lansky or Karnofsky Performance Score (KPS) of ≥ 70% at the time of entry.
* Laboratory Studies:

  1. Platelet count ≥ 125,000 per microliter prior to biopsy. Platelets ≥ 100,000 per microliter prior to infusion;
  2. Prothrombin and Activated Partial Thromboplastin Times ≤ 1.2 x upper limit of normal (ULN) prior to biopsy;
  3. Positive serum anti-poliovirus titer ≥ 1:8 prior to biopsy;
  4. Creatinine ≤ 1.2 x ULN prior to biopsy;
  5. Total bilirubin, AST, ALT, alkaline phosphatase ≤ 2.5 x ULN prior to biopsy;
  6. Neutrophil count ≥ 1000 per microliter prior to biopsy;
  7. Hemoglobin ≥ 9 gm/dl prior to biopsy (can be transfused).
* The patient must have received a boost immunization with trivalent inactivated IPOL™ (Sanofi-Pasteur) ≥ 1 week prior to administration of the study agent.
* At the time of biopsy, prior to administration of virus, the presence of recurrent tumor must be confirmed by histopathological analysis.
* A signed informed consent form approved by the Duke University Institutional Review Board (IRB) will be required for patient enrollment into the study. Patients (if 18 years old) or their parent(s) or guardian(s) must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study. All children will have to provide assent to the study.
* Able to undergo brain MRI with and without contrast without requiring general anesthesia.

Exclusion Criteria:

* Pregnant or breast-feeding. Female patients of child-bearing potential or female sexual partners (who are of child-bearing potential) of male patients must use at least one of the following methods of medically acceptable contraceptives: approved hormonal contraceptives (such as birth control pills, patches, implants or infusions), an intrauterine device (IUD), or a barrier method of contraception (such as a condom or diaphragm) used ith spermicide. Because all patients are required to have a boost immunization of trivalent inactivated IPOL™, there should be no risk of transmission of a mother to her fetus after receiving intracranial PVSRIPO. As such, patients who become pregnant after receiving PVSRIPO will continue to be monitored in the same manner, i.e. per protocol, unless the assessment is contra-indicated during pregnancy. Partners who become pregnant will sign a Pregnant Partner Information Form and information regarding the pregnancy and its outcome may be collected.
* Patients with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeon.
* Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F).
* Patients with known immunosuppressive disease or known human immunodeficiency virus infection.
* Patients with unstable or severe intercurrent medical conditions such as severe heart (New York Heart Association Class 3 or 4) or lung (FEV1 < 50%) disease, uncontrolled diabetes mellitus.
* Patients with allergy to human serum albumin.
* Current or history of anaphylactic reaction to gadolinium.
* A history of neurological complications due to past PV infection would imply previous virus replication in the CNS. Based on animal studies, previous exposure to poliovirus administered intracerebrally can reduce subsequent virus replication in the CNS.
* Patients who have not recovered from the toxic effects of prior chemo- and/or radiation therapy. Guidelines for this recovery period are dependent upon the specific therapeutic agent being used:

  1. Patients who are less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 consecutive scans with disease progression or histopathologic confirmation of recurrent tumor.
  2. Patients who have received chemotherapy or bevacizumab ≤ 4 weeks [except for nitrosourea (6 weeks) or metronomic dosed chemotherapy such as daily etoposide or cyclophosphamide (1 week)] prior to starting the study drug unless patients have recovered from side effects of such therapy.
  3. Patients who have received immunotherapy ≤ 4 weeks prior to starting the study drug unless patients have recovered from side effects of such therapy.
* Patients with neoplastic lesions in the brainstem, cerebellum, spinal cord, intraventricular tumors, pituitary tumors, leptomeningeal disease, or other locations at the discretion of the treating neurosurgeon.
* Patients with a diagnosis of agammaglobulinemia, that is:

  1. Undetectable anti-tetanus toxoid IgG
  2. Known history of agammaglobulinemia
* Patients who are on dexamethasone receiving > 4 mg/day in the two weeks prior to admission for intra-cerebral delivery of PVSRIPO or who demonstrate worsening steroid myopathy.
* Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darell Bigner, MD, PhD, Study Director — Istari Oncology, Inc.; Daniel Landi, MD, Principal Investigator — Duke University; Eric Thompson, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barkley A, Butler E, Park C, Friedman A, Landi D, Ashley DM, Bigner D, Bernstock JD, Friedman GK, Johnston JM, Thompson EM. The safety and accuracy of intratumoral catheter placement to infuse viral immunotherapies in children with malignant brain tumors: a multi-institutional study. J Neurosurg Pediatr. 2024 Jan 12;33(4):359-366. doi: 10.3171/2023.12.PEDS23404. Print 2024 Apr 1. PMID 38215438
- [Derived] Thompson EM, Landi D, Brown MC, Friedman HS, McLendon R, Herndon JE 2nd, Buckley E, Bolognesi DP, Lipp E, Schroeder K, Becher OJ, Friedman AH, McKay Z, Walter A, Threatt S, Jaggers D, Desjardins A, Gromeier M, Bigner DD, Ashley DM. Recombinant polio-rhinovirus immunotherapy for recurrent paediatric high-grade glioma: a phase 1b trial. Lancet Child Adolesc Health. 2023 Jul;7(7):471-478. doi: 10.1016/S2352-4642(23)00031-7. Epub 2023 Mar 30. PMID 37004712
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — http://www.cancer.duke.edu/btc/
- See also: The Preston Robert Tisch Brain Tumor Center at Duke Pediatric Program — http://tischbraintumorcenter.duke.edu/pediatrics

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants Treated: All participants received a single lerapolturev infusion.
Period: Overall Study
Arm/Group | All Participants Treated
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants Treated: All participants received a single open-label infusion of lerapolturev
Arm/Group | All Participants Treated
Number analyzed (Participants) | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 16.5 [11.0 to 18.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Unacceptable Toxicity
Description: Percentage of participants with unacceptable toxicity during the 14-day period post-PVSRIPO treatment
Time Frame: 14 days after treatment with PVSRIPO
Measure: Number; unit: percentage of participants
Arm/Group | All Participants Treated
Number analyzed (Participants) | 8
percentage of participants | 0

2. Primary Outcome: Percentage of Participants Requiring Low-dose Bevacizumab or Steroid
Description: The percentage of participants requiring low-dose bevcizumab or steroid due to an inflammatory reaction secondary to an immune response to lerapolturev treatment
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | All Participants Treated
Number analyzed (Participants) | 8
percentage of participants | 50

3. Secondary Outcome: Overall Survival
Description: Estimation of overall survival calculated at the time between lerapolturev infusion and death or last follow-up if the participant is alive using the Kaplan-Meier method
Time Frame: up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Participants Treated
Number analyzed (Participants) | 8
months | 4.1 [1.2 to 10.1]

ADVERSE EVENTS:
Time Frame: All adverse events were collected up to 1 year; all-cause mortality was assessed for up to 2 years
Arm/Group | All Participants Treated
All-Cause Mortality (participants affected / at risk) | 7/8
Serious Adverse Events (participants affected / at risk) | 5/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants Treated (N=8)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants Treated (N=8)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Fatigue (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (6)
Memory impairment (Nervous system disorders) | 2 (2)
Metabolism and nutrition disorders - other, specify (Metabolism and nutrition disorders) | 1 (1) — Night sweats
Nervous system disorders - other (Nervous system disorders) | 3 (5)
Papilledema (Eye disorders) | 1 (1)
Pyramidal tract syndrome (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03043391/Prot_SAP_000.pdf